CLINICAL TRIAL: NCT01184885
Title: A Pilot Study of Hyperfractionated Cyclophosphamide, Vincristine, Doxorubicin, and Dexamethasone (Hyper-CVAD) With Sirolimus for the Treatment of Adult Acute Lymphoblastic Leukemia and Aggressive Lymphoid Malignancies
Brief Title: A Pilot Study to Determine the Safety and Tolerability of Sirolimus Given With Hyper-CVAD Chemotherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09G.474; 2009-35 (Other: CCRRC); JT 1505 (Other: JeffTrial Number)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Lymphoid Malignancies (New or Relapsed); Acute Lymphoblastic Leukemia; Burkitt Lymphoma; Lymphoblastic Lymphoma; Mantle Cell Lymphoma; Adult T-cell Leukemia/Lymphoma
Keywords: hyperCVAD; rapamycin; lymphoid malignancies; lymphoblastic leukemia; B and T cell; philadelphia chromosome negative; burkitt lymphoma; burkitt-type lymphoma; lymphoblastic lymphoma; mantle cell lymphoma; adult t cell leukemia; adult t cell lymphoma
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — CVAD protocol; Cyclophosphamide; Vincristine; Doxorubicin; Methotrexate; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hyper-CVAD and Sirolimus (Experimental): Hyper-CVAD and Sirolimus
  Interventions: Drug: Hyper-CVAD; Drug: Sirolimus

INTERVENTIONS:
Drug: Hyper-CVAD — * Cycle A: Cyclophosphamide 300mg/m2 every 12 hours on days 3-5; Vincristine 2mg/day on days 6 and 13; Doxorubicin 50mg/m2 on day 6; Decadron 40mg/ day po on days 3-6 and 13-16; Methotrexate 12mg IT on day 4; Ara-C 100mg IT on day 9.
  * Cycle B: Methotrexate 1000mg/m2 on day 3; Leucovorin 50mg every 6 hours starting 24 hours from the beginning of the MTX infusion until MTX levels are < 0.1 umol/L; Ara-C 3000mg/m2 every 12 hours on days 4 and 5; Methotrexate 12mg IT on day 4; Ara-C 100mg IT on day 9.
  * Rituximab (if given) will be 375 mg/m2 on Days 3 and 13 of Cycle A and on Days 4 and 9 of cycle B, for a total of 8 doses over the first 4 courses.
  Other Names: Cytoxan; Endoxan; Neosar; Procytox; Revimmune; Cytophosphane; Oncovin; Leurocristine; Adriamycin; Hydroxydaunorubicin; MTX; Amethopterin
Drug: Sirolimus — Sirolimus loading dose of 12mg on day 1 followed by a single daily dose of 4 mg/ day on days 2 through 7 (Cycle A) and on days 2 through 6 (Cycle B)
  Other Names: Rapamycin

SUMMARY:
This is a pilot study, assessing the feasibility, safety and toxicity of an mTOR (mammalian target of Rapamycin) inhibitor (MTI), rapamycin, when administered with HyperCVAD (Hyperfractionated Cyclophosphamide, Vincristine, Doxorubicine and Dexamethasone), with an ultimate goal to perform a phase II study to evaluate response rates and survival in adults with Acute Lymphoblastic Leukemia (ALL) and aggressive lymphoid malignancies.

DETAILED DESCRIPTION:
The primary objective of this trial is to characterize the feasibility, safety and tolerability of therapy with Hyper-CVAD and Rapamycin in adults with ALL and other aggressive lymphoid malignancies.

This study will evaluate the effectiveness of Rapamycin given in combination with Hyper-CVAD during A treatment cycles, and Methotrexate and Cytarabine in B treatment cycles. Both cycles will also contain the drug Rituximab if the patient has a B cell type of leukemia or lymphoma.

This combination of drugs are being studied to determine whether or not these drugs will have an effect in treating this disease.

Current therapeutic regimens for induction of remission in ALL are broadly similar. There is no single best regimen for induction therapy. The hyper-CVAD regimen is of particular interest because it does not include asparaginase as part of the therapeutic regimen and the results of induction are similar to other published regimens.

The HyperCVAD regimen with or without rituximab is also an accepted induction regimen for lymphoblastic lymphoma, Burkitt and Burkitt like lymphoma, Mantle Cell Lymphoma, and ALL in the elderly. The regimen has also been used as a salvage regimen in patients with the above diagnoses who have relapsed after another induction regimen.

This trial will add a novel agent, an mTOR inhibitor (MTI), rapamycin, to act synergistically with the HyperCVAD regimen. This is a pilot study, assessing the feasibility, safety and toxicity of this regimen, with an ultimate goal to perform a phase II study to evaluate response rates and survival.

This is a pilot study of the Hyper-CVAD regimen with Rapamycin for the treatment of adults with acute lymphoblastic leukemia or other aggressive lymphoid malignancies. The standard Hyper-CVAD regimen will be used, with the addition of the investigational agent, Rapamycin. Hyper-CVAD alone is one of the current standard induction and salvage regimens used to treat ALL and other aggressive lymphoid malignancies.

Subjects included will have either de novo, relapsed, or refractory ALL or another aggressive lymphoid malignancy.

Chemotherapy will consist of 4 'A' cycles alternating with 4 'B' cycles, every 21 days, or as count recovery allows (at least 14 days apart) as follows: 1A; 1B; 2A; 2B, 3A; 3B; 4A; 4B. This is dependent on white blood cell count recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of one of the following lymphoid malignancies (new or relapsed):

   * Acute Lymphoblastic Leukemia (B and T cell, Philadelphia Chromosome Negative)
   * Burkitt Lymphoma
   * Burkitt - type Lymphoma
   * Lymphoblastic Lymphoma
   * Mantle Cell Lymphoma
   * Adult T cell Leukemia/ lymphoma
2. Patients must be >18 years old
3. Patients must have an ECOG performance status of 0 or 1(see attachment 1).
4. Patients must have a life expectancy of at least 4 weeks.
5. Patients must be able to consume oral medication.
6. Patients must have completed any radiotherapy four weeks prior to study entry, 0-2 weeks for local palliative XRT (small port).
7. Patients must have recovered from the toxic effects of any prior chemotherapy to < grade 2 (except alopecia).
8. Required initial laboratory values: Creatinine < or = 2.0mg/dL; total or direct bilirubin < or = 1.5mg/dL (if not due to the leukemia or lymphoma itself); SGPT(ALT) < or = 3xULN; glucose <200 mg/dL, negative pregnancy test for women with child-bearing potential.
9. Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
10. Patients may have had a prior stem cell transplant (autologous or allogeneic), however they may not have active GvHD, nor be on any immunosuppression

Exclusion Criteria:

1. Patients must not be receiving any chemotherapy agents (except Hydroxyurea)
2. Intrathecal ARA-C and intrathecal methotrexate are permissible (as they are not systemic and only isolated to the central nervous system).
3. Patients must not be receiving growth factors, except for erythropoietin.
4. Patients with a current second malignancy requiring systemic therapy, other than non-melanoma skin cancers, are not eligible.
5. Patients with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, myocardial infarction within the past 6 months or serious uncontrolled cardiac arrhythmia are not eligible.
6. Patients taking any of the following drugs while on-study are not eligible:

   1. Carbamazepine (e.g. Tegretol)
   2. Rifabutin (e.g. Mycobutin)
   3. Rifampin (e.g. Rifadin)
   4. Rifapentine (e.g. Priftin)
   5. St. John's Wort- may decrease the effects of sirolimus by decreasing the amount of sirolimus in the body
   6. Clarithromycin (e.g. Biaxin)
   7. Cyclosporin e.g. (Neorla or Sandimmune)
   8. Diltiazem (e.g. Cardizem)
   9. Erythromycin (e.g. Akne-Mycin, Ery-Tab)
   10. Itraconazole (e.g. Sporanox)
   11. Ketoconazole (e.g. Nizoral)
   12. Telithromycin (e.g. Ketek)
   13. Verapamil (e.g. Calan SR, Isoptin, Verelan)
   14. Voriconazole (e.g. VFEND) - May increase the effects of sirolimus by increasing the amount of this medicine in the body. [Cannot be taken within 72 hours prior to or subsequent to receiving rapamycin, but may be taken prior to or after the above time period]
   15. Tacrolimus (e.g. Prograf) - May cause liver transplant rejection or serious side effects in patients on sirolimus.
7. Patients with known HIV positivity or AIDS-related illness are not eligible.
8. Patients with other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study are ineligible.
9. Patients must not have evidence of cerebellar dysfunction or prior history of cerebellar dysfunction with Ara-C administration.
10. Patients must not have received any investigational agents within 30 days of study entry.
11. Patients must not be pregnant or breastfeeding. Pregnancy tests must be obtained for all females of child-bearing potential. Pregnant or lactating patients are ineligible for this study due to the unknown human fetal or teratogenic toxicities of rapamycin. Males or females of reproductive age may not participate unless they have agreed to use an effective contraceptive method.
12. Patients who have uncontrolled infection are not eligible. Patients must have any active infections under control. Fungal disease must be stable for at least 2 weeks before study entry. Patients with bacteremia must have documented negative blood cultures prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyper-CVAD and Sirolimus: Hyper-CVAD and Sirolimus
  Hyper-CVAD : - Cycle A: Cyclophosphamide 300mg/m2 every 12 hours on days 3-5; Vincristine 2mg/day on days 6 and 13; Doxorubicin 50mg/m2 on day 6; Decadron 40mg/ day po on days 3-6 and 13-16; Methotrexate 12mg IT on day 4; Ara-C 100mg IT on day 9.
  * Cycle B: Methotrexate 1000mg/m2 on day 3; Leucovorin 50mg every 6 hours starting 24 hours from the beginning of the MTX infusion until MTX levels are < 0.1 umol/L; Ara-C 3000mg/m2 every 12 hours on days 4 and 5; Methotrexate 12mg IT on day 4; Ara-C 100mg IT on day 9.
  * Rituximab (if given) will be 375 mg/m2 on Days 3 and 13 of Cycle A and on Days 4 and 9 of cycle B, for a total of 8 doses over the first 4 courses.
  Sirolimus : Sirolimus loading dose of 12mg on day 1 followed by a single daily dose of 4 mg/ day on days 2 through 7 (Cycle A) and on days 2 through 6 (Cycle B)
Period: Overall Study
Arm/Group | Hyper-CVAD and Sirolimus
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyper-CVAD and Sirolimus
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.68 (18.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Count Recovery That Allows for Starting a Phase II Study to Evaluate Response Rates and Survival
Description: This will be assessed by evaluating the tolerability of this regimen compared to historical controls who received Hyper-CVAD or Hyper-CVAD/ Rituximab regimens. The treatment will be designated feasible for an individual subject if in 80% of chemotherapy cycles the subject has count recovery that allows for starting the subsequent cycle by Day 28. Count recovery is defined as ANC (absolute neutrophil count) of > 0.5 x 10^9/L and platelet count > 50 x 10^9/L.
  Hyper-CVAD/Rapamycin will be deemed acceptable if it is feasible to administer in 80% or more of subjects.
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- Hyper-CVAD and Sirolimus: Hyper-CVAD and Sirolimus
  Hyper-CVAD : - Cycle A: Cyclophosphamide 300mg/m^2 every 12 hours on days 3-5; Vincristine 2mg/day on days 6 and 13; Doxorubicin 50mg/m^2 on day 6; Decadron 40mg/day po on days 3-6 and 13-16; Methotrexate 12mg IT on day 4; Ara-C 100mg IT on day 9.
  * Cycle B: Methotrexate 1000mg/m^2 on day 3; Leucovorin 50mg every 6 hours starting 24 hours from the beginning of the MTX infusion until MTX levels are < 0.1 umol/L; Ara-C 3000mg/m^2 every 12 hours on days 4 and 5; Methotrexate 12mg IT on day 4; Ara-C 100mg IT on day 9.
  * Rituximab (if given) will be 375 mg/m^2 on Days 3 and 13 of Cycle A and on Days 4 and 9 of cycle B, for a total of 8 doses over the first 4 courses.
  Sirolimus : Sirolimus loading dose of 12mg on day 1 followed by a single daily dose of 4 mg/day on days 2 through 7 (Cycle A) and on days 2 through 6 (Cycle B)
Arm/Group | Hyper-CVAD and Sirolimus
Number analyzed (Participants) | 7
participants | 7

2. Secondary Outcome: Induction Mortality
Description: Induction mortality. Hyper-CVAD/ Rapamycin will be considered acceptable if induction mortality does not exceed 31% in patients older than 60, or 15% in those younger than 60
Time Frame: 18 months
Reporting Status: Not Posted

3. Secondary Outcome: Complete Response
Description: To describe response rates to hyper-CVAD and sirolimus in adults with ALL and other aggressive lymphoid malignancies.
  Bone marrow (<5% blasts) with adequate bone marrow cellularity, no evidence of circulating blasts or extramedullary disease and normalization of peripheral blood counts except for platelets (neutrophil count =1,000/µL).
Time Frame: Every 21 days or as count recovery allows (at least 14 days apart) up to 24 weeks
Measure: Number; unit: participants
Arm/Group | Hyper-CVAD and Sirolimus
Number analyzed (Participants) | 7
participants | 4

ADVERSE EVENTS:
Arm/Group | Hyper-CVAD and Sirolimus
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyper-CVAD and Sirolimus (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (8)
Infection (Infections and infestations) | 2 (2)
Edema (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Speech impairment (General disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 2 (2)
Gram negative sepsis (Immune system disorders) | 1 (1)
Face pain (General disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic shock (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyper-CVAD and Sirolimus (N=7)
Shoulder pain (General disorders) | 1 (1)
Abdominal pain (General disorders) | 4 (5)
Weight gain (General disorders) | 2 (2)
Edema (Skin and subcutaneous tissue disorders) | 5 (10)
Fatigue (General disorders) | 7 (15)
Constipation (General disorders) | 2 (4)
Extremity swelling (General disorders) | 1 (1)
Itching (General disorders) | 4 (4)
Weakness (General disorders) | 7 (10)
Bad taste in mouth (General disorders) | 1 (1)
Nightmares (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (11)
Blood in stool (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Weight loss (General disorders) | 2 (3)
Sweats (General disorders) | 4 (7)
Chest pain (General disorders) | 4 (6)
Opacified left maxillary sinus (General disorders) | 1 (1)
Back pain (General disorders) | 4 (4)
Sinusitis (General disorders) | 1 (1)
Numbness/tingling (Nervous system disorders) | 3 (4)
Muscle pain/tightness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutropenic fever (General disorders) | 3 (5)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Chills (General disorders) | 5 (9)
Nausea (General disorders) | 6 (11)
Abdominal ascites (General disorders) | 1 (1)
Gingivitis (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Insomnia (General disorders) | 4 (4)
Cough (General disorders) | 4 (7)
Nocturia (Renal and urinary disorders) | 3 (3)
Stiff neck (General disorders) | 2 (2)
Congestion (General disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Fever (General disorders) | 5 (9)
Gastric reflux (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (12)
Vomiting (General disorders) | 4 (5)
Blurred vision (Eye disorders) | 1 (1)
Post nasal drip (General disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (2)
Nosebleed (General disorders) | 4 (6)
Hypoxia (General disorders) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lightheadedness (General disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Stomach upset (Gastrointestinal disorders) | 2 (2)
Abscess (Skin and subcutaneous tissue disorders) | 2 (2)
Infection (Infections and infestations) | 3 (4)
Neuropathy (Nervous system disorders) | 4 (6)
Alopecia (General disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Poor appetite (General disorders) | 5 (5)
Positive blood culture (Blood and lymphatic system disorders) | 2 (3)
Low platelets (Blood and lymphatic system disorders) | 1 (1)
Tooth problem (General disorders) | 2 (2)
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Pulse oxygen dropped (Blood and lymphatic system disorders) | 1 (1)
Mouth sores (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Blood and lymphatic system disorders) | 2 (3)
Facial flushing (Skin and subcutaneous tissue disorders) | 2 (2)
Confusion (Psychiatric disorders) | 3 (4)
Headache (General disorders) | 4 (9)
Speech impairment (General disorders) | 1 (1)
Throat pain (General disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Double vision (Eye disorders) | 1 (1)
Unable to move right eye (Eye disorders) | 1 (1)
Lower abductor pain (General disorders) | 1 (1)
Trouble sleeping (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (9)
Taste alteration (General disorders) | 1 (1)
Hip pain (General disorders) | 1 (1)
Cold (General disorders) | 1 (1)
Groin nodule (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus congestion (General disorders) | 2 (2)
Hyperpigmented circumscribed areas on scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Respiratory infection (Infections and infestations) | 1 (1)
Bone pain (General disorders) | 3 (3)
Sore throat (General disorders) | 2 (2)
Wrist pain (General disorders) | 1 (1)
Ankle pain (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3)
Eye conjunctival redness (Eye disorders) | 1 (1)
Gas/bloating (Gastrointestinal disorders) | 2 (2)
Agitation (General disorders) | 2 (2)
Mood alteration (Psychiatric disorders) | 2 (2)
Psychosis (Psychiatric disorders) | 2 (2)
Rigidity (General disorders) | 1 (1)
Catatonia (Psychiatric disorders) | 1 (1)
Difficulty swallowing (General disorders) | 1 (1)
Dizziness (General disorders) | 2 (2)
Puffy face (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Swollen ankles (General disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Mouth/throat discomfort (General disorders) | 1 (1)
Rectal pain (General disorders) | 1 (1)
Abnormal gait (General disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Jaw pain (General disorders) | 2 (2)
Leg pain (General disorders) | 1 (1)
Soft tissue swelling (General disorders) | 1 (1)
Irregular heartbeat (Cardiac disorders) | 1 (1)
Achiness (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Sinus headache (General disorders) | 1 (1)
Soreness of tongue (General disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Stomach pain (General disorders) | 1 (1)
Mucositis (General disorders) | 1 (1)
Bleeding from PICC site (General disorders) | 1 (1)
Choreiform movement (Nervous system disorders) | 1 (1)
Transfusion reaction (General disorders) | 1 (1)
Decreased urine output (Renal and urinary disorders) | 1 (1)
Lactic acidosis (Blood and lymphatic system disorders) | 1 (1)
Elevated bilirubin (General disorders) | 1 (2)
Eyes appear uncoordinated (Eye disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Bleeding from IV site (General disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Autodiuresis/polyuria (Renal and urinary disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Anal incontinence (General disorders) | 1 (1)
Increased troponins (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Jaundice (Skin and subcutaneous tissue disorders) | 1 (1)
Oral bleeding (General disorders) | 1 (1)
Rib pain (General disorders) | 1 (1)
Decreased bowel sounds (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Absent breath sounds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Volume overload (General disorders) | 1 (1)
Abdominal tenderness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes